CLINICAL TRIAL: NCT02282059
Title: A Multi Center, Prospective, Non Interventional (NI) Study of the Safety and Efficacy of Sunitinib in Chinese Patients With Progressive Advanced or Metastatic Well Differentiated Unresectable Pancreatic Neuroendocrine Tumors
Brief Title: The Safety And Efficacy Of Sunitinib In Chinese Patients With Progressive Advanced Or Metastatic Well-Differentiated Unresectable Pancreatic Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181215
Record Dates: First submitted 2014-10-15; First posted 2014-11-04 (Estimated); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Neuroendocrine Tumors
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sunitinib group: patients with progressive, unresectable, advanced or metastatic well-differentiated pNET
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — subjects will be enrolled to receive at least one dose of sunitinib orally at 37.5 mg once a day on a continuous daily dosing regimen (CDD) or dosage modification is based on daily clinic practice

SUMMARY:
This study is a multi-center, prospective, non-interventional (NI) study evaluating the safety and efficacy of sunitinib in Chinese patients with progressive, unresectable, advanced or metastatic well-differentiated, pancreatic neuroendocrine tumors(pNET). 100 adults with progressive advanced or metastatic well-differentiated unresectable pNET will be recruited in China hospitals. Each subject will be followed up overall survival (OS) time or the date of withdrawal and subjects who remain alive after study completion will have their OS time censored on the last date known to be alive. Eligible subjects will be enrolled to receive at least one dose of sunitinib orally at 37.5 mg once a day on a continuous daily dosing regimen (CDD) or dosage modification is based on daily clinic practice. Subjects will be treated until disease progress, unacceptable toxicity, withdrawal from the study at their own request, or until the final analysis for the study is performed. The NI study will capture observations that will be used for evaluating the safety profile of sunitinib, including: subject demographics, medical history and medications. Safety assessments, treatment data and any other laboratory examination results, which were done according to routine clinical practice, will be collected at all visits.

DETAILED DESCRIPTION:
The sunitinib non-interventional (NI) study is a real world observational study which represents the usual and customary treatment of patients and being proposed to collect data systematically and to assess the safety and efficacy in Chinese patients with progressive, unresectable, advanced or metastatic well-differentiated, pancreatic neuroendocrine tumors.It is designed and conducted to meet CFDA post-marketing commitments. non-probability sample

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing to follow up visits within current clinical practice.
* Histologically or cytologically proven diagnosis of well-differentiated pancreatic neuroendocrine tumors (according to WHO 2000 classification)
* Unresectable (as assessed by the investigator) or metastatic disease documented on a scan
* A minimum age of 18 years

Exclusion Criteria:

* Patients with poorly-differentiated pancreatic neuroendocrine tumors (according to WHO 2000 classification)
* Patients who have received at least one dosage of sunitinib treatment prior to signing informed consent form will be excluded from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Chinese adult with progressive advanced or metastatic well-differentiated unresectable pancreatic neuroendocrine tumors is the target population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- China (24):
  - Oncology Department, The Second Affiliated Hospital of Anhui Medical University, Hefei, An'hui
  - Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated Tumour Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Eastern Theater General Hospital,QinHuai District Medical Area, Nanjing, Jiangsu
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command/Hepatobiliary Surgery Department, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Digestive surgery Department, The First Affiliated Hospital, The Fourth Military Medical University, Xi'an, Shannxi
  - The First Affiliated Hospital，Air Force Medical University, Xi'an, Shannxi
  - Air Force Medical University, Xi’an, Shanxi
  - West China Hospital of Sichuan University/Hepatobiliary Pancreatic Surgery, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Oncology department, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Fifth Medical Center of PLA General Hospital, Beijing
  - The PLA of 307 Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University General Hospital/General Surgery, Tianjin
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181215&StudyName=A%20Multi-center%2C%20Prospective%2C%20Non-interventional%20%28NI%29%20Study%20Of%20The%20Safety%20And%20Efficacy%20Of%20Sunitinib%20In%20Chinese%20Patients%20With%20Progressive%20Advanced%20Or%20Metastatic%20Well-differentiated%20Unresectable%20Pancreatic%20Neuroendocrine%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 participants were enrolled and assigned to the study treatment, and 99 participants were treated.
Groups:
- Sunitinib (Not Taken): Sunitinib (Not Taken) were the participants with progressive, unresectable, advanced or metastatic well-differentiated pancreatic neuroendocrine tumors who would accept sunitinib therapy when signing informed consent.
- Sunitinib (Already Taken): Sunitinib (Already Taken) were the participants with progressive, unresectable, advanced or metastatic well-differentiated pancreatic neuroendocrine tumors who had already taken sunitinib within the past 6 months (26 weeks) when signing informed consent and would continue sunitinib therapy.
Period: Overall Study
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Started | 82 | 18
Treated (One participant (not taken sunitinib before) who had been assigned to the study treatment was not treated and therefore excluded from the study analysis.) | 81 | 18
Discontinued (Discontinued participants included those who completed minimum 5-year follow-up since they have been assigned to the study treatment.) | 82 | 18
Completed | 0 | 0
Not Completed | 82 | 18
Not completed — Other | 15 | 3
Not completed — Participant refused further follow-up | 8 | 4
Not completed — Lost to Follow-up | 19 | 3
Not completed — Death | 40 | 8

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants who took at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken) | Total
Number analyzed (Participants) | 81 | 18 | 99
Age, Continuous [Median (Full Range); unit: Years] | 52.0 [24 to 73] | 49.0 [21 to 75] | 51.0 [21 to 75]
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  18-44 years | 26 | 5 | 31
  45-64 years | 40 | 11 | 51
  >=65 years | 15 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 6 | 37
  Male | 50 | 12 | 62
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 81 | 18 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All Causalities and Treatment-related)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product. The event did not necessarily need to have a causal relationship with the product treatment or usage. A TEAE was defined as an event that emerged during treatment, having been absent pretreatment, or worsened relative to the pretreatment state.
Time Frame: From baseline up to 8 years
Population: The safety analysis population included all enrolled participants who took at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Participants
  All-causality TEAEs | 61 | 13
  Treatment-related TEAEs | 52 | 12

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) (All Causalities and Treatment-related)
Description: An SAE was any untoward medical occurrence in a participant administered a medicinal at any dose that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect.
Time Frame: From baseline up to 8 years
Population: The safety analysis population included all enrolled participants who took at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Participants
  All-causality SAEs | 11 | 5
  Treatment-related SAEs | 2 | 2

3. Primary Outcome: Number of Participants With Hematology/Chemistry/Urinalysis Laboratories of Baseline Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤2 at Baseline That Shifted to a Maximum CTCAE Grade 3 or 4
Description: Laboratory abnormalities assessment included: hematologic: hemoglobin, platelet count, white blood cell (WBC) count, neutrophile granulocyte count; non-hematologic: total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, gamma-glutamyl transferase (GGT), total protein, albumin, blood urea nitrogen (BUN), creatinine, uric acid, glucose, hypocalcemia, hyponatremia, hypophosphatemia, hypokalaemia.
Time Frame: From baseline up to 8 years
Population: The safety analysis population included all enrolled participants who took at least 1 dose of the study drug. Participants with missing first dosing date were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Participants
  Anemia (Grade 0 to Grade 3): number analyzed (Participants) | 68 | 16
  Anemia (Grade 0 to Grade 3) | 2 | 2
  Anemia (Grade 1 to Grade 3): number analyzed (Participants) | 68 | 16
  Anemia (Grade 1 to Grade 3) | 1 | 1
  Anemia (Grade 2 to Grade 3): number analyzed (Participants) | 68 | 16
  Anemia (Grade 2 to Grade 3) | 4 | 1
  Lymphocyte count decreased (Grade 0 to Grade 3): number analyzed (Participants) | 68 | 16
  Lymphocyte count decreased (Grade 0 to Grade 3) | 4 | 1
  Lymphocyte count decreased (Grade 1 to Grade 3): number analyzed (Participants) | 68 | 16
  Lymphocyte count decreased (Grade 1 to Grade 3) | 1 | 0
  Lymphocyte count decreased (Grade 2 to Grade 3): number analyzed (Participants) | 68 | 16
  Lymphocyte count decreased (Grade 2 to Grade 3) | 1 | 0
  Neutrophil count decreased (Grade 0 to Grade 3): number analyzed (Participants) | 68 | 16
  Neutrophil count decreased (Grade 0 to Grade 3) | 7 | 3
  Neutrophil count decreased (Grade 1 to Grade 3): number analyzed (Participants) | 68 | 16
  Neutrophil count decreased (Grade 1 to Grade 3) | 1 | 1
  Neutrophil count decreased (Grade 1 to Grade 4): number analyzed (Participants) | 68 | 16
  Neutrophil count decreased (Grade 1 to Grade 4) | 1 | 0
  Platelet count decreased (Grade 0 to Grade 3): number analyzed (Participants) | 68 | 16
  Platelet count decreased (Grade 0 to Grade 3) | 2 | 1
  Platelet count decreased (Grade 1 to Grade 3): number analyzed (Participants) | 68 | 16
  Platelet count decreased (Grade 1 to Grade 3) | 0 | 1
  Platelet count decreased (Grade 0 to Grade 4): number analyzed (Participants) | 68 | 16
  Platelet count decreased (Grade 0 to Grade 4) | 1 | 0
  Platelet count decreased (Grade 1 to Grade 4): number analyzed (Participants) | 68 | 16
  Platelet count decreased (Grade 1 to Grade 4) | 1 | 0
  WBC decreased (Grade 0 to Grade 3): number analyzed (Participants) | 67 | 16
  WBC decreased (Grade 0 to Grade 3) | 4 | 1
  WBC decreased (Grade 1 to Grade 3): number analyzed (Participants) | 67 | 16
  WBC decreased (Grade 1 to Grade 3) | 1 | 1
  WBC decreased (Grade 1 to Grade 4): number analyzed (Participants) | 67 | 16
  WBC decreased (Grade 1 to Grade 4) | 1 | 0
  ALT increased (Grade 0 to Grade 3): number analyzed (Participants) | 68 | 16
  ALT increased (Grade 0 to Grade 3) | 1 | 0
  ALT increased (Grade 1 to Grade 3): number analyzed (Participants) | 68 | 16
  ALT increased (Grade 1 to Grade 3) | 1 | 0
  ALT increased (Grade 2 to Grade 3): number analyzed (Participants) | 68 | 16
  ALT increased (Grade 2 to Grade 3) | 1 | 0
  Alkaline phosphatase increased (Grade 0 to Grade 3): number analyzed (Participants) | 67 | 16
  Alkaline phosphatase increased (Grade 0 to Grade 3) | 1 | 0
  Alkaline phosphatase increased (Grade 1 to Grade 3): number analyzed (Participants) | 67 | 16
  Alkaline phosphatase increased (Grade 1 to Grade 3) | 1 | 0
  AST increased (Grade 1 to Grade 3): number analyzed (Participants) | 68 | 16
  AST increased (Grade 1 to Grade 3) | 2 | 0
  Blood bilirubin increased (Grade 0 to Grade 3): number analyzed (Participants) | 68 | 16
  Blood bilirubin increased (Grade 0 to Grade 3) | 3 | 0
  Blood bilirubin increased (Grade 2 to Grade 3): number analyzed (Participants) | 68 | 16
  Blood bilirubin increased (Grade 2 to Grade 3) | 1 | 0
  GGT increased (Grade 1 to Grade 3): number analyzed (Participants) | 66 | 16
  GGT increased (Grade 1 to Grade 3) | 4 | 0
  GGT increased (Grade 2 to Grade 3): number analyzed (Participants) | 66 | 16
  GGT increased (Grade 2 to Grade 3) | 4 | 1
  GGT increased (Grade 0 to Grade 4): number analyzed (Participants) | 66 | 16
  GGT increased (Grade 0 to Grade 4) | 1 | 1
  Hyperglycemia (Garde 0 to Grade 3): number analyzed (Participants) | 62 | 14
  Hyperglycemia (Garde 0 to Grade 3) | 2 | 0
  Hypocalcemia (Garde 0 to Grade 3): number analyzed (Participants) | 56 | 11
  Hypocalcemia (Garde 0 to Grade 3) | 0 | 1
  Hypokalemia (Garde 0 to Grade 3): number analyzed (Participants) | 60 | 11
  Hypokalemia (Garde 0 to Grade 3) | 4 | 0
  Hypokalemia (Garde 2 to Grade 3): number analyzed (Participants) | 60 | 11
  Hypokalemia (Garde 2 to Grade 3) | 2 | 0
  Hypokalemia (Garde 2 to Grade 4): number analyzed (Participants) | 60 | 11
  Hypokalemia (Garde 2 to Grade 4) | 0 | 1
  Hyponatremia (Garde 0 to Grade 3): number analyzed (Participants) | 61 | 11
  Hyponatremia (Garde 0 to Grade 3) | 2 | 0
  Hypophosphatemia (Garde 0 to Grade 3): number analyzed (Participants) | 48 | 10
  Hypophosphatemia (Garde 0 to Grade 3) | 1 | 0
  Hypophosphatemia (Garde 2 to Grade 3): number analyzed (Participants) | 48 | 10
  Hypophosphatemia (Garde 2 to Grade 3) | 2 | 0

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Investigator assessed PFS according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.6. PFS was defined as the time from the start of sunitinib treatment to first document of objective tumor progression or death due to any cause, whichever occurred first. Progression was defined using RECIST v1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From baseline up to 8 years
Population: The analysis population included all participants who took at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Months | 10.4 [4.6 to NA] — Upper limit of the 95% Confidence Interval was not estimable due to an insufficient number of participants with events. | 25.5 [8.3 to 42.7]

5. Secondary Outcome: Progression-Free Survival by Clinical Judgment
Description: PFS by clinical judgment was defined as the time from the start of sunitinib treatment to first document of objective tumor progression, or first time tumor progression diagnosed by investigator based on clinical judgment, or death due to any cause, whichever occurred first. Progression was defined using RECIST v1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From baseline up to 8 years
Population: The analysis population included all participants who took at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Months | 10.4 [4.6 to 27.6] | 42.7 [3.8 to 42.7]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of sunitinib treatment to documentation of death due to any cause.
Time Frame: From baseline up to 8 years
Population: The analysis population included all participants who took at least 1 dose of the study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Months | 46.2 [30.0 to 77.9] | NA [14.7 to NA] — Upper limit of the 95% Confidence Interval was not estimable due to an insufficient number of participants with events.

7. Secondary Outcome: Five-Year Survival Rate
Description: Five-year survival rate was defined as the proportion of participants who stayed alive till after 5 years from the start of sunitinib treatment.
Time Frame: From baseline up to 8 years
Population: The analysis population included all participants who took at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken)
Number analyzed (Participants) | 81 | 18
Proportion of participants | 0.478 [0.352 to 0.594] | 0.504 [0.249 to 0.714]

ADVERSE EVENTS:
Time Frame: From baseline up to 8 years
Groups:
- Total: (=sum per row)
Arm/Group | Sunitinib (Not Taken) | Sunitinib (Already Taken) | Total
All-Cause Mortality (participants affected / at risk) | 40/81 | 8/18 | 48/99
Serious Adverse Events (participants affected / at risk) | 11/81 | 5/18 | 16/99
Other Adverse Events (participants affected / at risk) | 55/81 | 13/18 | 68/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (Not Taken) (N=81) | Sunitinib (Already Taken) (N=18) | Total (N=99)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Death (General disorders) | 1 | 0 | 1 — 2 cases were reported with AE term as Death.The AE term for 1 participant was "unknown cause of death".Death reason for the other one was disease progression.So data here was updated to 1.The other one was added to SAE of Disease progression below.
Disease progression (General disorders) | 2 | 1 | 3
Oedema peripheral (General disorders) | 0 | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 3 | 0 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (Not Taken) (N=81) | Sunitinib (Already Taken) (N=18) | Total (N=99)
Anaemia (Blood and lymphatic system disorders) | 19 | 6 | 25
Myelosuppression (Blood and lymphatic system disorders) | 3 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 7 | 5 | 12
Eyelid oedema (Eye disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 7 | 3 | 10
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 4
Ascites (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 11
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 1 | 7
Vomiting (Gastrointestinal disorders) | 9 | 3 | 12
Chest pain (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 1 | 2
Oedema peripheral (General disorders) | 3 | 1 | 4
Pyrexia (General disorders) | 6 | 0 | 6
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 11 | 3 | 14
Aspartate aminotransferase increased (Investigations) | 11 | 5 | 16
Blood albumin decreased (Investigations) | 3 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 7 | 2 | 9
Blood bilirubin increased (Investigations) | 5 | 1 | 6
Blood calcium decreased (Investigations) | 0 | 2 | 2
Blood creatinine increased (Investigations) | 5 | 0 | 5
Blood glucose increased (Investigations) | 3 | 1 | 4
Blood potassium decreased (Investigations) | 1 | 2 | 3
Blood urea increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 1
Fibrin D dimer increased (Investigations) | 2 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 7 | 5 | 12
Haemoglobin decreased (Investigations) | 4 | 3 | 7
Lymphocyte count decreased (Investigations) | 2 | 4 | 6
Neutrophil count decreased (Investigations) | 25 | 7 | 32
Platelet count decreased (Investigations) | 26 | 6 | 32
Protein total decreased (Investigations) | 1 | 1 | 2
Red blood cell count decreased (Investigations) | 1 | 1 | 2
White blood cell count decreased (Investigations) | 27 | 9 | 36
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 1 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 1 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 10 | 0 | 10
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 1 | 8
Portal vein embolisation (Surgical and medical procedures) | 0 | 1 | 1
Hypertension (Vascular disorders) | 8 | 1 | 9

LIMITATIONS AND CAVEATS:
Due to the real world nature of this study, heterogeneity of clinical judgment and clinical practice may exist which may include but it not limited to the following: timing of imaging/laboratory testing, different measurement techniques/standards for judging tumor change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02282059/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02282059/SAP_001.pdf